CLINICAL TRIAL: NCT05218382
Title: A Randomized Study on Use of Virtual Reality Technology for Pain Relief in Transvaginal Oocyte Retrieval Under Conscious Sedation
Brief Title: Pain Relief Using VR in Oocyte Retreival
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Ernest Hung-Yu Ng, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TUGOR-VR
Record Dates: First submitted 2021-12-18; First posted 2022-02-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Infertility; Pain
Keywords: VR; IVF; oocyte retrieval; pain levels
MeSH Terms: conditions — Infertility; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled superiority trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding of the participants is not possible due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): The participants will have the the virtual reality headset with immersive virtual reality.
  Interventions: Device: Virtual reality
- Placeob group (Placebo Comparator): The participants will have the virtual reality headset put on but blank screen.
  Interventions: Device: No virtual reality

INTERVENTIONS:
Device: Virtual reality — immersive virtual reality technology
  Arms: VR group
Device: No virtual reality — Virtual reality with blank screen
  Arms: Placeob group

SUMMARY:
Title: A randomized study on use of virtual reality technology for pain relief in transvaginal oocyte retrieval under conscious sedation Objectives: The study is to evaluate the effectiveness of virtual reality (VR) in pain relief during transvaginal ultrasound-guided oocyte retrieval (TUGOR) under conscious sedation Hypothesis to be tested: VR can reduce the pain level during TUGOR. Design and subjects: This is a randomized study on additional use of VR during TUGOR. A total of 160 women undergoing oocyte retrieval on both ovaries will be recruited and randomized to one of the following groups: active and placebo groups. Those with known allergy to pethidine, diazepam or local anaesthetics; and history of claustrophobia/ susceptible to motion sickness will be excluded.

Instruments: Immersive VR Interventions: All received women will receive the standard conscious sedation with 25mg IV pethidine and 5mg IV diazepam; and paracervical block of 10ml 1% lignocaine. VR headset will be put on for every woman. It will only be switched on for the active VR group but not the placebo VR group.

Main outcome measures: The primary outcome measure is the maximal abdominal pain levels during TUGOR measured by a 100mm linear visual analogue scale prior. Secondary outcome measures include the pain of vaginal puncture and the abdominal pain four hours after the procedure prior to discharge from hospital.

Data analysis and expected results: Data will be analysed on intention to treat basis and per protocol. Demographic features of the study groups will be compared. Chi-square test or Fisher's exact test will be used for categorical variables. Mann-Whitney U test will be used to compare the continuous variables between groups. P values of <0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
Introduction Transvaginal ultrasound guided oocyte retrieval is an essential process in in-vitro fertilization. The procedure lasts for around 10-15 minutes and is considered as a painful procedure. Different modalities of pain relief methods are used including paracervical blocks(1-3), conscious sedation (4, 5), spinal anaesthesia and general anaesthesia (6). Conscious sedation with anaesthesia was the commonly chosen method in assisted reproduction technology centers; as it enhances a faster post-procedure recovery and less anaesthetic risks as compared with general anaesthesia.

Recently, the use of immersive virtual reality technology has been applied in pain control in different medical fields especially in paediatrics, oncology and burn patients (7, 8). It provides a distraction from the acute pain during procedures and its effectiveness has been shown in meta-analysis (9, 10). In gynaecology, use of VR can significantly reduce the pain in ambulatory hysteroscopy (score 6.0 versus 3.7, p = 0.0009) (11). Another group of investigators also initiated a study on VR as pain relief in hysterosalpingogram (12). While, there is no study evaluating the use of VR in transvaginal oocyte retrieval.

In view of that, the aim of this study is to evaluate the effectiveness of VR in pain relief during transvaginal oocyte retrieval under conscious sedation.

Trial objectives and hypothesis:

The objective is to evaluate the effectiveness of VR in pain relief during transvaginal oocyte retrieval using conscious sedation.

Hypothesis VR can reduce the pain experienced during transvaginal oocyte retrieval using conscious sedation.

Trial design This is a randomized study on additional use of VR during transvaginal oocyte retrieval using conscious sedation. All subjects will receive the standard conscious sedation with 25mg IV pethidine and 5mg IV diazepam; and paracervical local anaesthetic 10ml 1% lignocaine. In addition, they will be randomized to receive immersive VR or not.

Treatment of subjects:

Women undergoing in-vitro fertilization at Department of Obstetrics and Gynaecology of Queen Mary Hospital will be assessed for eligibility. Eligible women will be recruited for the study and informed written consent will be obtained after written and oral information.

Eligible women recruited will be randomly assigned on the day of oocyte retrieval according to a computer-generated randomization list into one of the following two groups.

1. VR group - The women will receive Immersive VR.
2. Placebo group - They will have the VR headset put on but blank screen. Blinding of the subjects is not possible due to the nature of the intervention.

Ovarian stimulation and oocyte retrieval will be performed according to departmental Standard Operating Procedures. The VR headset will be put on prior to oocyte retrieval and it will be turned on in the VR group only. The headset will be cleansed with wipes after each use. Disposable hygiene masks will be used below the headset.

25mg Pethidine and 5mg Diazepam will be given intravenously. The blood pressure and pulse of the women are checked after the drug administration and the oxygen saturation is monitored continuously throughout the procedure. 10ml 1% lignocaine is injected to the paracervical region by the operating surgeon with a 21-gauge needle after cleansing of the vagina and cervix with chlorhexidine. Under transvaginal ultrasound guidance, a 16-gauge ovum aspiration needle is introduced. Aspiration of follicles without flushing is performed with a suction pressure of 100mmHg.

Assessment of anxiety Shortly after hospital admission in the morning, women will complete the state-trait anxiety inventory (STAI) questionnaire before oocyte retrieval to assess their trait and state anxiety.

Assessment of pain levels and sedation levels The women will be asked to rate according to a 100mm linear visual analogue scale prior to start of procedure, within 5 minutes after the procedure and four hours after the procedure prior to discharge from hospital.

They will be asked to rate:

* The anticipated pain during the procedure
* The worst pain during the procedure

The surgeon will score the sedation level of the women according to the scale described by Ramsay et al., at the end of the operation. Level 1: Patient anxious and agitated or restless or both; Level 2: Patient co-operative, orientated, and tranquil; Level 3: Patient responsive to commands only; Level 4: Asleep and a brisk response to loud auditory stimulus; Level 5: Asleep and a sluggish response to loud auditory stimulus; Level 6: Asleep and no response to loud auditory stimulus.

Any adverse effects experienced such as (nausea, vomiting, dizziness, drowsiness will be recorded.

They will be asked to complete the client satisfaction questionnaire before discharge.

Basic demographic data will be collected including age, indication of infertility, number of oocytes obtained, and duration of procedure.

No extra follow-up visits will be arranged solely for the study unless considered necessary by the investigators.

ELIGIBILITY:
Inclusion Criteria:

* - women aged > 18 years and <43 years

  * understand Chinese
  * undergoing transvaginal oocyte retrieval on both sides

Exclusion Criteria:

* Had known allergy to pethidine, diazepam or local anaesthetics
* Had oocyte retrieval performed on one ovary only
* History of claustrophobia/ susceptible to motion sickness

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile women undergoing oocyte retrieval
Enrollment: 160 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Pain levels | Day 0
  maximal pain level during oocyte retrieval experienced by the participants measured by visual analog scale from 0-100 (maximum); higher levels mean mean painful

SECONDARY OUTCOMES:
level of unpleasantness | Day 0
  level of unpleasantness during oocyte retrieval (nil, mild, moderate and severe)
client satisfaction questionnaire score | Day 0
  scoring of client satisfaction questionnaire from 10 (minimum) to 40 (maximum); higher scores mean higher satisfaction
Ongoing pregnancy rate | 10 weeks
  Pregnancy rate at 8-10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ng, MD, Study Director — The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
No similar studies in this area
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available upon publication of the study and be available for 10 years.
Access Criteria: any reasonable request

REFERENCES:
- [Result] Ng EH, Miao B, Ho PC. A randomized double-blind study to compare the effectiveness of three different doses of lignocaine used in paracervical block during oocyte retrieval. J Assist Reprod Genet. 2003 Jan;20(1):8-12. doi: 10.1023/a:1021202604049. PMID 12645862
- [Result] Ng EH, Tang OS, Chui DK, Ho PC. Comparison of two different doses of lignocaine used in paracervical block during oocyte collection in an IVF programme. Hum Reprod. 2000 Oct;15(10):2148-51. doi: 10.1093/humrep/15.10.2148. PMID 11006189
- [Result] Ng EH, Tang OS, Chui DK, Ho PC. A prospective, randomized, double-blind and placebo-controlled study to assess the efficacy of paracervical block in the pain relief during egg collection in IVF. Hum Reprod. 1999 Nov;14(11):2783-7. doi: 10.1093/humrep/14.11.2783. PMID 10548622
- [Result] Kwan I, Wang R, Pearce E, Bhattacharya S. Pain relief for women undergoing oocyte retrieval for assisted reproduction. Cochrane Database Syst Rev. 2018 May 15;5(5):CD004829. doi: 10.1002/14651858.CD004829.pub4. PMID 29761478
- [Result] Lai SF, Lam MT, Li HWR, Ng EHY. A randomized double-blinded non-inferiority trial comparing fentanyl and midazolam with pethidine and diazepam for pain relief during oocyte retrieval. Reprod Biomed Online. 2020 May;40(5):653-660. doi: 10.1016/j.rbmo.2020.01.021. Epub 2020 Jan 31. PMID 32299734
- [Result] Roest I, Buisman ETIA, van der Steeg JW, Koks CAM. Different methods of pain relief for IVF and ICSI oocyte retrieval - A Dutch survey. Eur J Obstet Gynecol Reprod Biol X. 2019 Jun 15;4:100065. doi: 10.1016/j.eurox.2019.100065. eCollection 2019 Oct. PMID 31517299
- [Result] Dunn J, Yeo E, Moghaddampour P, Chau B, Humbert S. Virtual and augmented reality in the treatment of phantom limb pain: A literature review. NeuroRehabilitation. 2017;40(4):595-601. doi: 10.3233/NRE-171447. PMID 28211829
- [Result] Indovina P, Barone D, Gallo L, Chirico A, De Pietro G, Giordano A. Virtual Reality as a Distraction Intervention to Relieve Pain and Distress During Medical Procedures: A Comprehensive Literature Review. Clin J Pain. 2018 Sep;34(9):858-877. doi: 10.1097/AJP.0000000000000599. PMID 29485536
- [Result] Mallari B, Spaeth EK, Goh H, Boyd BS. Virtual reality as an analgesic for acute and chronic pain in adults: a systematic review and meta-analysis. J Pain Res. 2019 Jul 3;12:2053-2085. doi: 10.2147/JPR.S200498. eCollection 2019. PMID 31308733
- [Result] Ahmad M, Bani Mohammad E, Anshasi HA. Virtual Reality Technology for Pain and Anxiety Management among Patients with Cancer: A Systematic Review. Pain Manag Nurs. 2020 Dec;21(6):601-607. doi: 10.1016/j.pmn.2020.04.002. Epub 2020 May 15. PMID 32423641
- [Result] Deo N, Khan KS, Mak J, Allotey J, Gonzalez Carreras FJ, Fusari G, Benn J. Virtual reality for acute pain in outpatient hysteroscopy: a randomised controlled trial. BJOG. 2021 Jan;128(1):87-95. doi: 10.1111/1471-0528.16377. Epub 2020 Jul 22. PMID 32575151
- [Result] Wang YL, Gao HX, Wang JS, Wang JH, Bo L, Zhang TT, Dai YL, Gao LL, Liu Q, Zhang JJ, Cai JM, Yu JQ, Li YX. Immersive virtual reality as analgesia for women during hysterosalpingography: study protocol for a randomized controlled trial. Trials. 2020 Jan 20;21(1):102. doi: 10.1186/s13063-019-4023-y. PMID 31959220
- [Derived] Ng CSM, Tong PYW, Wong E, Cheng HHY, Ko JKY, Li RHW, Ng EHY. Randomized controlled study on the use of virtual reality for pain relief in oocyte retrieval under transvaginal ultrasound guidance using paracervical block and conscious sedation. Hum Reprod. 2025 Dec 1;40(12):2310-2317. doi: 10.1093/humrep/deaf188. PMID 40974211